CLINICAL TRIAL: NCT06898762
Title: Creation of a National Multicenter Platform for the Study of Inflammatory Myocardial Disease: Pre-MYO Cohort
Acronym: PREMYO
Status: Recruiting | Type: Observational
Sponsor: Fundacion para la Formacion e Investigacion Sanitarias de la Region de Murcia (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-5-2-HCUVA
Record Dates: First submitted 2025-03-21; First posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Myocarditis Acute; Inflammatory Cardiomyopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: characterization of a large national cohort of patients with suspected myocarditis or inflammatory cardiomyopathy. — characterization of a large national cohort of patients with suspected myocarditis or inflammatory cardiomyopathy.

SUMMARY:
The objectives of this project are: 1) to comprehensively characterize a large national cohort of patients with suspected myocarditis, their clinical phenotype, care management, blood and imaging biomarkers, epidemiological, environmental and genetic data; 2) to retrospectively validate the accuracy of the new hsa-RNA-Chr8:96 biomarker for the diagnosis of myocarditis compared to conventional diagnosis; 3) to identify acquired and inherited mutations, and their interaction with the environment, which explain the susceptibility to myocarditis, its severity and response to treatment; 4) to study the lower incidence in women and the influence of age, considering socio-health and genetic factors.

DETAILED DESCRIPTION:
The primary endpoint of the study will be the characterization of a broad national cohort of patients with suspected myocarditis or inflammatory cardiomyopathy. The secondary endpoints of the study will be (A) individual susceptibility to developing myocarditis or inflammatory cardiomyopathy, 1) identifying acquired and inherited genetic variants, and 2) from the persistence of gender, age, and socioenvironmental conditions; and (B) studying the correlation between the final diagnosis of myocarditis and the hsa-miR-Chr8:96 marker.

ELIGIBILITY:
Inclusion Criteria:

• Presence of at least one compatible symptom and at least one objective finding in diagnostic tests (Figure 2), according to the consensus document of the European Society of Cardiology (1):

A. Clinical presentation:

* Acute chest pain: pericardial or pseudo-ischemic.
* Dyspnea on exertion or at rest for up to 3 months.
* Dyspnea on exertion or at rest for 3 months - 1 year.
* Unexplained palpitations / arrhythmias, sudden death recovered.
* Unexplained cardiogenic shock.

B. Findings in complementary tests:

* ECG: new onset AV block, new onset bundle branch block, ST segment elevation/depression, T wave inversion
* Elevation of TnI/TnT
* Segmental or global contractility alterations not explained by other causes
* Positive Lake Louise criteria in cardiac MRI (13) (Annex III Figure S1) • Patients who have given their informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with clinical suspicion of myocarditis or inflammatory cardiomyopathy will be included, based on the presence of compatible clinical findings.
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2023-04-09 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
characterization of a large national cohort of patients with suspected myocarditis or inflammatory cardiomyopathy. | Up to 3 years
  Subjects will be recruited during an emergency room visit or within their usual clinical practice among those patients who meet the criteria for participation in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Domingo Pascual Figal, MD, Principal Investigator — HCUVA
Locations (1):
- HCUVA, Murcia, Murcia, Spain